CLINICAL TRIAL: NCT02083848
Title: Detection of Loco-regional Invasion of Cervical Cancer With 7 Tesla MRI (DETECT)
Brief Title: Detection of Loco-regional Invasion of Cervical Cancer With 7 Tesla MRI
Acronym: DETECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, W.B. Veldhuis, MD PhD, Radiologist, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL41056.041.13
Record Dates: First submitted 2014-03-04; First posted 2014-03-11 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Cervical Cancer
Keywords: Locoregional invasion; Stage IB1, IB2, IIA or IIB
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 7T MRI (Other): All subjects are entered into a single arm.
  Interventions: Other: 7T MRI

INTERVENTIONS:
Other: 7T MRI — Ultra high field magnetic resonance imaging

SUMMARY:
Background of the study: The accurate assessment of local cervical cancer spread (i.e. invasion) is of clinical importance for staging and treatment considerations. For example, if parametrial invasion is absent, radical surgery is the treatment of choice for tumors less than 4cm in diameter. However, if such invasion is present, the patient has become inoperable and (chemo)radiotherapy is warranted. Unfortunately, regular 1.5T MRI as a part of staging work-up has a limited accuracy for detecting loco-regional tumor invasion. Due to relatively frequent false-negative findings a risk of understaging and under-treatment occurs. For such cases adjuvant treatments with (chemo)radiotherapy are indicated after the initial surgery, causing increased morbidity and treatment associated risks. For higher stages, with primary (chemo)radiotherapy, a more reliable MRI based delineation of local tumor spread could enable individualized dose(volume) and field modifications.

Hypothesis/aim of the study: To develop and in vivo optimize T2w ultra high field (7T) MRI sequences, which use a combination of an endorectal and external coil, to image the (para)cervical area for assessment of the loco-regional tumor status in cervical cancer.

Study design: The proposed study is an investigator initiated, single center, prospective pilotstudy.

Study population: 20 patients with histological proven cervical cancer stage IB1, IB2, IIA of IIB will be included.

Primary study parameters/outcome of the study: Optimized T2w ultra high field (7T) MRI sequences of the (para)cervical area which allow qualitative assessment of the loco-regional invasion of cervical cancer.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven primary malignancy of the cervix uteri;
* FIGO stage IB1, IB2, IIA or IIB;
* ≥18 years;
* Written inform consent provided.

Exclusion Criteria:

* Contra-indications for MRI: Any non-removable electronic or ferromagnetic object present in the body; Pregnancy; Severe claustrophobia; Unable to lie still and completely horizontal for minimally 45 minutes;
* Body weight >150kg;
* Any type of neo-adjuvant chemo- and/or radiotherapy for cervical cancer;
* Uterine prolapse with C ≥ -6 cm (POP-Q).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Optimized T2w ultra high field (7T) MRI sequence of the (para)cervical area which allow qualitative assessment of the loco-regional invasion of cervical cancer. | Up to 2 years from study initiation
  This is a feasibility outcome (feasibility study). This pilot study does not aim to test diagnostic accuracy. The (feasibility) criteria when this 7T MRI protocol is deemed optimized are:
  * Successful depiction, at minimum, of the anatomy present in the inner pelvis (at the cervical level) in three orthogonal planes;
  * Sufficient T2w contrast in the created datasets for clinical diagnostic applicability. This includes sufficient T2w contrast within the cervix to be able to delineate its subanatomy (e.g. mucosa vs. fibrous tissue);
  * Absence of image distorting artefacts, which reduce the clinical diagnostic applicability, regardless of their cause;
  * The overall protocol does not exceed 45 minutes of scan time;
  * Reproducibility of the above mentioned criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob P Hoogendam, MD, Study Director — UMC Utrecht; Wouter B Veldhuis, MD PhD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands